CLINICAL TRIAL: NCT00595907
Title: Observational Study of Production of IFN-Gamma by Peripheral Lymphocytes in Response to Specific Antigens Before and After Treatment for Tuberculosis
Brief Title: Results of an Interferon-Gamma Release Assay After Treatment for Tuberculosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Jean-Paul Janssens, MD
Other Study IDs: Janssens1/2008
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Tuberculosis
Keywords: tuberculosis; interferon gamma release assays; treatment
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood lymphocytes cultured over-night; ELISPOT for detection of interferon-gamma production
Oversight: Data Monitoring Committee: Yes

SUMMARY:
New blood tests have become available to detect either latent or active tuberculosis. These tests - which according to the CDC can replace the tuberculin skin test - measure the production of gamma-interferon (a cytokine) by peripheral lymphocytes (white cells) when exposed to antigens which are highly specific of mycobacterium tuberculosis (the bacteria responsible for tuberculosis). Our hypothesis was that the production of gamma-interferon would be much higher at the beginning of treatment than at the end, and that decline in gamma-interferon secretion could be an indicator of clinical response to treatment.

DETAILED DESCRIPTION:
Patients either treated for active culture proven tuberculosis (TB) or having completed treatment during the preceding 6 months were recruited. Exclusion criteria were : HIV infection and previous TB. Interferon gamma release assay (T-SPOT.TB, Oxford Immunotec) was sampled during the 2 first weeks of treatment, at the end of treatment and 6 months later.

T-SPOT.TB was analysed qualitatively (pos/neg) and quantitatively (Spot forming units: SFU) to determine if there was a higher rate of negative tests at the end of treatment and 6 months after treatment than initially. Paired samples were analysed to compare SFU counts between beginning of treatment and end of treatment, and SFU counts between end of treatment and 6 months later.

Clinical response to treatment was recorded, as well as treatment failures and relapses.

ELIGIBILITY:
Inclusion Criteria:

* culture proven tuberculosis

Exclusion Criteria:

* age < 18
* prior tuberculosis
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients either at diagnosis of tuberculosis, under treatment for tuberculosis, or within 6 months after treatment completion
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2004-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Interferon gamma response to M. tuberculosis antigens by peripheral lymphocytes after treatment for tuberculosis | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, M.D., Principal Investigator — University Hospital, Geneva
Locations (1):
- Centre antituberculeux; Geneva University Hospital, Geneva, Geneva 14, Switzerland

REFERENCES:
- [Background] Janssens JP, Roux-Lombard P, Perneger T, Metzger M, Vivien R, Rochat T. Quantitative scoring of an interferon-gamma assay for differentiating active from latent tuberculosis. Eur Respir J. 2007 Oct;30(4):722-8. doi: 10.1183/09031936.00028507. Epub 2007 May 30. PMID 17537773
- [Derived] Bosshard V, Roux-Lombard P, Perneger T, Metzger M, Vivien R, Rochat T, Janssens JP. Do results of the T-SPOT.TB interferon-gamma release assay change after treatment of tuberculosis? Respir Med. 2009 Jan;103(1):30-4. doi: 10.1016/j.rmed.2008.09.012. Epub 2008 Nov 1. PMID 18977647